CLINICAL TRIAL: NCT06446986
Title: Dual Task Effect in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aynur Başaran, Proffessor Dr, MD, Karamanoğlu Mehmetbey University
Other Study IDs: 01-2024/06
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Scoliosis Idiopathic
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with adolescent idiopathic scoliosis
  Interventions: Other: Single and Dual-Task Timed Up and Go Test; Other: Single and Dual-Task Tandem Walking Test; Other: Simple Shoulder Test
- Control group: Age and sex matched healthy adolescent peers
  Interventions: Other: Single and Dual-Task Timed Up and Go Test; Other: Single and Dual-Task Tandem Walking Test; Other: Simple Shoulder Test

INTERVENTIONS:
Other: Single and Dual-Task Timed Up and Go Test — Timed Up and Go Test will be conducted. Then, for motor-motor dual-task evaluation, the test will be repeated while the subjects carry a tray containing 4 glasses of water without spilling the water. The time required to complete each test will be recorded in seconds.
Other: Single and Dual-Task Tandem Walking Test — The tandem walking test will be performed. Then, for cognitive-motor dual-task tandem walking test assessment, the test will be repeated while the subject completes one of 3 different cognitive tasks. These cognitive tasks used during dual-task trials will be switched between trials in an attempt to avoid a practice effect. The time required to complete each test will be recorded in seconds.
  The cognitive tasks are as follows:
  1. Counting down by six or seven from a randomly presented 2-digit number
  2. Counting backward the months starting from a randomly selected month
  3. Spelling a five-letter word backwards
Other: Simple Shoulder Test — Simple Shoulder Test contains 12 items and rates pain and function in patients with shoulder problems. Each item has two options and is scored either ''1 = yes'' or ''0 = no''. The total score ranges from 0 to 12. Higher scores indicate better physical functions.

SUMMARY:
The goal of this observational study is to evaluate the dual task and upper extremity disability in individuals with adolescent idiopathic scoliosis compared to healthy controls and to examine their relationship with clinical and radiological parameters in adolescent idiopathic scoliosis (AIS). The main questions it aims to answer are:

1. To compare dual task and upper extremity disability in individuals with AIS and healthy sex and age-matched healthy controls.
2. To analyze the relationship of dual-task and upper extremity disability in individuals with AIS with clinical and radiological parameters All participants' dual-task performance will be evaluated and they will answer the upper extremity disability survey. Besides, the study groups will be examined thoroughly and radiological parameters will be calculated to identify the clinical and radiological parameters that affect dual-task performance and upper extremity disability.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional deformity and sagittal plane changes are accompanied by coronal plane changes. As a result of spinal deformity, morphological changes occur in the trunk and rib cage, and the relationships between body parts are affected. Considering the anatomical proximity between the scapula and the rib cage, alteration of the shoulder and upper extremity functions as a consequence of the change in proximal orientation is expected.

On the other hand, maintaining postural control depends on the dynamic relationship between sensory information and motor output. Dual tasking is an experience-based neurophysiological process that requires a person to perform two tasks simultaneously. When a person has problems with the neurophysiological process, the performance of one or both functions is negatively affected.

This observational study aims to evaluate the dual task and upper extremity disability in individuals with adolescent idiopathic scoliosis compared to healthy controls and to examine their relationship with clinical and radiological parameters in AIS. All participants' dual-task performance will be evaluated and they will answer the upper extremity disability survey. Besides, the study groups will be examined thoroughly and radiological parameters will be calculated to identify the clinical and radiological parameters that affect dual-task performance and upper extremity disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Adolescent Idiopathic Scoliosis

Exclusion Criteria:

* Patients with complaints of neck, back, and shoulder pain
* Having a known neurological or systemic disease
* Having cognitive dysfunction that cannot cooperate with evaluations
* Having undergone musculoskeletal surgery or injury
* Extremity length difference of more than 1 cm
* Regular repetitive overhead shoulder movements related to professional or sports activities
* BMI >30 kg/m2

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescent Idiopathic Scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
The difference in seconds of the Single and Dual-Task Timed Up and Go Test between study and control groups | baseline
  Univariate statistical analyses will be performed to calculate the differences in seconds between the study group and control group.
The difference in seconds of the Single and Dual-Task Tandem Walking Test between study and control groups | baseline
  Univariate statistical analyses will be performed to calculate the differences in seconds between the study group and control group.
The difference of the Simple Shoulder Test scores between study and control groups | baseline
  Univariate statistical analyses will be performed to calculate the differences in the scores between the study group and control group.

SECONDARY OUTCOMES:
Multivariate analyses will be carried out with control variables | baseline
  Significant primary outcome measures will be controlled with:
  * Clinical parameters:
    * Scapular dyskinesia evaluation (present/absent)
    * Lateral scapular shift test (positive/negative)
    * TRACE score (Trunk Aesthetic Clinical Evaluation) (score ranges from 0 to12)
    * Thoracic expansion (cm)
  * Radiological parameters: Coronal plan:
    * Curve type (single, double major),
    * Location of curvature (Thoracic, thoracolumbar, lumbar),
    * Majör curve side (right/left),
    * Major curve Cobb angle (degrees),
    * Coronal balance (mm),
    * Apical vertebrae translation (mm),
    * Apical vertebrae rotation (Grade from 0 to 4),
    * Pelvic obliquity (degrees),
    * Radiographic shoulder height (mm),
  * Radiological parameters: Sagital plan
    * Torasik kyphosis Cobb angle (degrees),
    * Lumbar lordosis Cobb angle (degrees),
    * Sagittal balance (mm),
    * Pelvic tilt (degrees),
    * Sacral slope (degrees),
    * Pelvic incidence (degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Elif D Durmaz, Study Chair — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)